CLINICAL TRIAL: NCT06515990
Title: A Phase 1, Multicenter, Open-label, First-in-human, Dose Escalation and Expansion Study of DM005 in Patients With Advanced Solid Tumors
Brief Title: A Study of DM005 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Doma Biopharmaceutical（Suzhou）Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DM005001
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Solid Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (Experimental): 0.5mg/kg
  Interventions: Drug: DM005
- Dose Level 2 (Experimental): ≤1 mg/kg
  Interventions: Drug: DM005
- Dose Level 3 (Experimental): ≤2 mg/kg
  Interventions: Drug: DM005
- Dose Level 4 (Experimental): ≤4 mg/kg
  Interventions: Drug: DM005
- Dose Level 5 (Experimental): ≤6 mg/kg
  Interventions: Drug: DM005
- Dose Level 6 (Experimental): ≤8 mg/kg
  Interventions: Drug: DM005

INTERVENTIONS:
Drug: DM005 — An IV infusion of DM005 will be administrated approximately 30-60 min on D1 once Q3W.

SUMMARY:
The goal of this clinical trial is to find out about the safety, efficacy, and tolerability of DM005 for patients with the advanced solid tumors. DM005 is an experimental drug which is not approved by health authorities for the treatment of advanced solid tumors. For each participant, there will be a screening period of up to 28 days, a treatment period consisting of 21-day cycles, an end of treatment (EOT) Visit (+7 days), and a Follow-up Visit at 30 days (±7 days) after the EOT Visit.

Participants with advanced solid malignant tumors will be treated with DM005 on Day 1 of each cycle (every 3 weeks, Q3W). An initial dose of DM005 will be infused intravenously (IV) into each participant for approximately 60 minutes (±10) on Cycle1 Day 1. If there is no infusion-related reaction (IRR) during or after the initial dose, with the Investigator's confirmation and supervision, the subsequent dosing of DM005 in the following cycles maybe infused IV for approximately 30 minutes ( ±5). A 21-day observation period (Cycle 1) will then occur, at the end of which all relevant safety data will be reviewed.

DETAILED DESCRIPTION:
This first-in-human (FIH), multicenter, open-label, dose escalation and dose expansion study is to evaluate the safety, preliminary efficacy and pharmacokinetic (PK) characteristics of DM005 monotherapy in participants with advanced solid tumors.

DM005, a bispecific ADC developed using fully human antibodies with a common light chain, which targets c-MET and EGFR.

Subjects with solid malignant tumors will be treated with DM005 on Day 1 once Q3W (dose adjustments may be required depending on the safety profile and PK data of each dose

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criteria for both Parts

  1. Participants must have the ability to understand and willingness to sign a written informed consent document.
  2. Participants who have pathologically or cytologically documented metastatic/advanced NSCLC, gastroesophageal cancer, CRC, HCC, pancreatic cancer, or HNSCC, not curable with standard local therapies (i.e., surgery and/or radiation) and have progressed on standard therapy, or intolerant to standard therapy.
  3. Participants must be ≥18 years of age on the day of signing the informed consent form (ICF).
  4. Participants must have an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 2.
  5. Has a life expectancy ≥3 months.
  6. Has measurable disease based on response evaluation criteria in solid tumors (RECIST) version 1.1.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. Participants have another active invasive malignancy within 5 years, with the following exceptions and notes:

     * History of noninvasive malignancy, such as cervical cancer in situ, in situ melanoma, or ductal carcinoma in situ of the breast that is in complete remission years after treatment with curative intent is allowed.
     * Malignancies with a negligible risk of metastasis or death (such as adequately treated basal or squamous cell skin cancer and localized prostate cancer).
  2. Current or history of hematologic malignancy.
  3. Anticancer therapy (chemotherapy, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, or other anti-cancer therapies, except for hormones for hypothyroidism or estrogen replacement therapy, anti-estrogen analogs, agonists required to suppress serum testosterone levels) within 28 days or 5 half-lives, whichever is shorter, prior to the first study dose. Radiotherapy with a wide field of radiation within 28 days, or radiotherapy with a limited field of radiation for palliation within 14 days of the first study dose. Major surgery, other than diagnostic surgery, within 4 weeks of the first study dose.
  4. Primary central nervous system (CNS) malignancies or CNS metastases. Individuals with brain metastases can be enrolled only if treated, non-progressive brain metastases and off high-dose steroids (>20 mg prednisone or equivalent) for at least 4 weeks.
  5. Presence of bulky disease (defined as any single mass >7 cm in its greatest dimension). Individuals with a mass >7 cm, but otherwise eligible, may be considered for enrollment after discussion and approval with the medical monitor.
  6. Has an uncontrolled infection requiring IV injection of antibiotics, antivirals, or antifungals.
  7. Has clinically significant corneal disease.
  8. Has a corrected QT interval (QTcF) prolongation to >470 ms (for both genders) based on average of the Screening triplicate 12-lead ECG determinations; no concomitant medications that would prolong the QT interval; no known family history of long QT syndrome.
  9. Left ventricular ejection fraction (LVEF) <50% by either an echocardiogram (ECHO) or a multigated acquisition (MUGA) scan within 28 days before first dose of the study drug.
  10. Known active hepatitis B (HBV) or hepatitis C (HCV) infection. Chronic carriers of HBV infection (HBsAg-positive, undetectable HBV DNA or HBV DNA ≤2500 copies/ml or 500 IU/ml) receive prophylactic treatment during the study can be enrolled. Participants with a history of HCV infection have completed curative antiviral treatment and HCV viral load below the limit of quantification and HCV antibody positive but HCV ribonucleic acid (RNA) negative due to prior treatment or natural resolution should be eligible.
  11. Known human immunodeficiency virus (HIV) infection which is not well controlled. participants should be tested for HIV prior to enrollment if required by local regulations or institutional review board (IRB)/ethics committee. All the following criteria are required to define an HIV infection (positive HIV1/2 antibodies test) that is well controlled: HIV viral load <400 copies/mL, CD4+ T-cell counts ≥350 cells/μL, no history of acquired immunodeficiency syndrome [AIDS])-defining opportunistic infection within the past 12 months, and stable viral load for at least 4 weeks on same anti-HIV retroviral medications.
  12. Participants from endemic area will be specifically screened for tuberculosis. Participants with active tuberculosis are excluded. Participants who have received bacille Calmette-Guerin (BCG) vaccination may have a false positive result in the purified protein derivative (PPD) skin test. These participants are eligible if they have a negative Interferon Gamma Release Assay (IGRA).
  13. Has received a live vaccine within 30 days prior to the first dose of study drug.
  14. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia and anemia) not yet resolved to NCI-CTCAE version 5.0, ≤Grade 1 or baseline. Note: Participants may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to enrollment/randomization and managed with the standard treatment) that the Investigator deems related to previous anticancer therapy, following discussion with the Sponsor's medical monitor, such as the following: Grade 2 chemotherapy-induced neuropathy, hypothyroidism, hyperglycemia.
  15. Females who are pregnant or lactating or who intend to become pregnant during participation in the study.
  16. Participants who are of reproductive potential refuse to use effective methods of birth control during participation of the study and within 7 months for female (and 4 months for male) after the last dose administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) of DM005 | 12 months
  Incidence of DLTs of DM005 will be determined. A dose-limiting toxicity (DLT) was defined as grade 3 neurological toxicities (e.g. chemical meningitis) or other grade 4 toxicity.
Maximum tolerated dose (MTD) for DM005 | 12 months
  The MTD of DM005 will be determined. The MTD was defined as the dose where 0/3 or 1/6 patients experienced a DLT with at least two patients encountering DLT at the higher dose.

SECONDARY OUTCOMES:
The MTD of DM005 will be determined. The MTD was defined as the dose where 0/3 or 1/6 patients experienced a DLT with at least two patients encountering DLT at the higher dose. | 12 months
  Area under the plasma concentration-time curve from time zero extrapolated to infinity, calculated by linear up/log down trapezoidal summation.
Maximum (peak) plasma concentration (Cmax, ng/mL) | 12 months
  Maximum concentration, obtained directly from the observed concentration versus time data.
Time to maximum (peak) concentration (Tmax, h) | 12 months
  Time to Cmax
Trough concentration (Ctrough, ng/mL) | 12 months
  The lowest plasma concentration reached before the next dose.
Objective response rate (ORR) | 12 months
  ORR is defined as the number of patients with at least a confirmed complete response (CR) or partial response (PR), based on the best objective response values while on treatment using RECIST version 1.1

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University Hospital, North Ryde, New South Wales
  - ICON Cancer Center, South Brisbane, Queensland